CLINICAL TRIAL: NCT03766191
Title: The Relation of Genetic Factors, Food Cues, and Self-Regulation With Excess Consumption and Adiposity in Children
Brief Title: Genetic Predisposition to Food Cue Reactivity in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Dartmouth College (Other)
Responsible Party: Principal Investigator, Diane Gilbert-Diamond, Associate Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: D19064; 1R01HD092604 (NIH)
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Childhood Obesity
Keywords: Obesity; Cue Reactivity; Genetics; Self Regulation; fMRI; Children; Eating in the Absence of Hunger
MeSH Terms: conditions — Pediatric Obesity; Obesity; Self-Control

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Food Ads and fMRI (Active Comparator): Exposure to food ads during an fMRI scan
  Interventions: Behavioral: Food Ads
- Non-Food Ads and fMRI (Sham Comparator): Exposure to non-food ads during an fMRI scan
  Interventions: Other: Non-food Ads
- Food Ads and TV show (Active Comparator): Exposure to food ads embedded in an age-appropriate TV program
  Interventions: Behavioral: Food Ads
- Non-Food Ads and TV show (Sham Comparator): Exposure to non-food ads embedded in an age-appropriate TV program
  Interventions: Other: Non-food Ads

INTERVENTIONS:
Behavioral: Food Ads — Exposure to foods ads embedded in an age-appropriate TV program
  Arms: Food Ads and TV show; Food Ads and fMRI
Other: Non-food Ads — Exposure to non-food ads embedded in an age-appropriate TV program
  Arms: Non-Food Ads and TV show; Non-Food Ads and fMRI

SUMMARY:
This study assesses the associations between genetic factors, food-cue-related neural reactivity, self-regulatory capacity, eating in the absence of hunger (EAH), and adiposity gain in children.

DETAILED DESCRIPTION:
The investigators will assess the associations between genetic factors, food-cue-related neural reactivity, eating in the absence of hunger (EAH) in response to food cues, and adiposity gain in children. They will also determine whether self-regulatory capacity modifies these associations. The genetic factors explored specifically include FTO, MC4R, polymorphisms in genes involved in dopaminergic pathways, and a composite genetic risk score built from genome-wide obesity-related loci.

[3/14/2020]: Study recruitment temporarily halted due to the COVID-19 pandemic

ELIGIBILITY:
Inclusion Criteria:

* English fluency
* Willingness to participate in all study visits

Exclusion Criteria:

* Relevant food allergies or dietary restrictions
* Metal in or on the body
* Claustrophobia
* Psychiatric and neurological disorders
* Relative in the study
* Appetite- or attention-altering medications or disorders

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Food-cue-related neural activity | Baseline
  Activation in brain reward regions in response to food vs. non-food cues, as measured by differences in the blood-oxygen-level dependent response during fMRI scans. Investigators will examine associations between polymorphisms in FTO, MC4R, as well as a genetic risk score with the differential neural activity.
Food-cue-related Eating in the Absence of Hunger (EAH) | Baseline, 2 weeks, 4 weeks
  Difference in kcals consumed in response to food vs. non-food cue exposure in the behavioral sessions. Investigators will examine how differential neural activity in response to food vs. non-food cues will relate to EAH. Investigators will also assess whether self-regulatory capacity diminishes this association between differential neural activity and EAH.
Change in BMI | Baseline, 1-year followup
  Difference between BMI z-score according to the Center for DiseaSe Control 2000 Growth Reference Curves assessed at baseline and follow-up. Investigators will assess the associations between genetic factors (polymorphisms in FTO, MC4R; and a genetic obesity risk score), food-cue-related neural activity and EAH with change in BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Gilbert-Diamond, ScD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Daniels SR, Arnett DK, Eckel RH, Gidding SS, Hayman LL, Kumanyika S, Robinson TN, Scott BJ, St Jeor S, Williams CL. Overweight in children and adolescents: pathophysiology, consequences, prevention, and treatment. Circulation. 2005 Apr 19;111(15):1999-2012. doi: 10.1161/01.CIR.0000161369.71722.10. PMID 15837955
- [Background] Freedman DS, Mei Z, Srinivasan SR, Berenson GS, Dietz WH. Cardiovascular risk factors and excess adiposity among overweight children and adolescents: the Bogalusa Heart Study. J Pediatr. 2007 Jan;150(1):12-17.e2. doi: 10.1016/j.jpeds.2006.08.042. PMID 17188605
- [Background] Dietz WH. Overweight in childhood and adolescence. N Engl J Med. 2004 Feb 26;350(9):855-7. doi: 10.1056/NEJMp048008. No abstract available. PMID 14985480
- [Background] Guo SS, Chumlea WC. Tracking of body mass index in children in relation to overweight in adulthood. Am J Clin Nutr. 1999 Jul;70(1):145S-148S. doi: 10.1093/ajcn/70.1.145s. PMID 10393162
- [Background] Guyenet SJ, Schwartz MW. Clinical review: Regulation of food intake, energy balance, and body fat mass: implications for the pathogenesis and treatment of obesity. J Clin Endocrinol Metab. 2012 Mar;97(3):745-55. doi: 10.1210/jc.2011-2525. Epub 2012 Jan 11. PMID 22238401
- [Background] Lutter M, Nestler EJ. Homeostatic and hedonic signals interact in the regulation of food intake. J Nutr. 2009 Mar;139(3):629-32. doi: 10.3945/jn.108.097618. Epub 2009 Jan 28. PMID 19176746
- [Background] Boswell RG, Kober H. Food cue reactivity and craving predict eating and weight gain: a meta-analytic review. Obes Rev. 2016 Feb;17(2):159-77. doi: 10.1111/obr.12354. Epub 2015 Dec 8. PMID 26644270
- [Background] Gilbert-Diamond D, Emond JA, Lansigan RK, Rapuano KM, Kelley WM, Heatherton TF, Sargent JD. Television food advertisement exposure and FTO rs9939609 genotype in relation to excess consumption in children. Int J Obes (Lond). 2017 Jan;41(1):23-29. doi: 10.1038/ijo.2016.163. Epub 2016 Sep 22. PMID 27654143
- [Background] Baumeister RF, Heatherton TF. Self-Regulation Failure: An Overview. Psychological Inquiry. 2009;7(1):1-15. doi:10.1207/s15327965pli0701_1.
- [Background] Heatherton TF, Wagner DD. Cognitive neuroscience of self-regulation failure. Trends Cogn Sci. 2011 Mar;15(3):132-9. doi: 10.1016/j.tics.2010.12.005. Epub 2011 Jan 26. PMID 21273114
- [Background] Muraven M, Baumeister RF, Tice DM. Longitudinal improvement of self-regulation through practice: building self-control strength through repeated exercise. J Soc Psychol. 1999 Aug;139(4):446-57. doi: 10.1080/00224549909598404. PMID 10457761
- [Background] Gailliot MT, Plant EA, Butz DA, Baumeister RF. Increasing self-regulatory strength can reduce the depleting effect of suppressing stereotypes. Pers Soc Psychol Bull. 2007 Feb;33(2):281-94. doi: 10.1177/0146167206296101. PMID 17259587
- [Background] Costanzo PR, Woody EZ. Domain-specific parenting styles and their impact on the child's development of particular deviance: the example of obesity proneness. Journal of social and clinical psychology. 1985;3(4):425-445.
- [Background] Fisher JO, Birch LL. Restricting access to palatable foods affects children's behavioral response, food selection, and intake. Am J Clin Nutr. 1999 Jun;69(6):1264-72. doi: 10.1093/ajcn/69.6.1264. PMID 10357749
- [Background] Birch LL, Fisher JO, Davison KK. Learning to overeat: maternal use of restrictive feeding practices promotes girls' eating in the absence of hunger. Am J Clin Nutr. 2003 Aug;78(2):215-20. doi: 10.1093/ajcn/78.2.215. PMID 12885700
- [Background] Santini F, Maffei M, Pelosini C, Salvetti G, Scartabelli G, Pinchera A. Melanocortin-4 receptor mutations in obesity. Adv Clin Chem. 2009;48:95-109. PMID 19803416
- [Background] Lim BK, Huang KW, Grueter BA, Rothwell PE, Malenka RC. Anhedonia requires MC4R-mediated synaptic adaptations in nucleus accumbens. Nature. 2012 Jul 11;487(7406):183-9. doi: 10.1038/nature11160. PMID 22785313
- [Background] Cui H, Mason BL, Lee C, Nishi A, Elmquist JK, Lutter M. Melanocortin 4 receptor signaling in dopamine 1 receptor neurons is required for procedural memory learning. Physiol Behav. 2012 May 15;106(2):201-10. doi: 10.1016/j.physbeh.2012.01.025. Epub 2012 Feb 9. PMID 22342812
- [Background] Srisai D, Gillum MP, Panaro BL, Zhang XM, Kotchabhakdi N, Shulman GI, Ellacott KL, Cone RD. Characterization of the hyperphagic response to dietary fat in the MC4R knockout mouse. Endocrinology. 2011 Mar;152(3):890-902. doi: 10.1210/en.2010-0716. Epub 2011 Jan 14. PMID 21239438
- [Background] Yilmaz Z, Davis C, Loxton NJ, Kaplan AS, Levitan RD, Carter JC, Kennedy JL. Association between MC4R rs17782313 polymorphism and overeating behaviors. Int J Obes (Lond). 2015 Jan;39(1):114-20. doi: 10.1038/ijo.2014.79. Epub 2014 May 14. PMID 24827639
- [Background] Han JC, Lawlor DA, Kimm SY. Childhood obesity. Lancet. 2010 May 15;375(9727):1737-48. doi: 10.1016/S0140-6736(10)60171-7. Epub 2010 May 5. PMID 20451244
- [Background] Biro FM, Wien M. Childhood obesity and adult morbidities. Am J Clin Nutr. 2010 May;91(5):1499S-1505S. doi: 10.3945/ajcn.2010.28701B. Epub 2010 Mar 24. PMID 20335542
- [Background] Whitaker RC, Wright JA, Pepe MS, Seidel KD, Dietz WH. Predicting obesity in young adulthood from childhood and parental obesity. N Engl J Med. 1997 Sep 25;337(13):869-73. doi: 10.1056/NEJM199709253371301. PMID 9302300
- [Background] Serdula MK, Ivery D, Coates RJ, Freedman DS, Williamson DF, Byers T. Do obese children become obese adults? A review of the literature. Prev Med. 1993 Mar;22(2):167-77. doi: 10.1006/pmed.1993.1014. PMID 8483856
- [Background] Clinical guidelines on the identification, evaluation, and treatment of overweight and obesity in adults: executive summary. Expert Panel on the Identification, Evaluation, and Treatment of Overweight in Adults. Am J Clin Nutr. 1998 Oct;68(4):899-917. doi: 10.1093/ajcn/68.4.899. No abstract available. PMID 9771869
- [Background] Collins FS, Varmus H. A new initiative on precision medicine. N Engl J Med. 2015 Feb 26;372(9):793-5. doi: 10.1056/NEJMp1500523. Epub 2015 Jan 30. PMID 25635347
- [Background] Gillman MW, Hammond RA. Precision Treatment and Precision Prevention: Integrating "Below and Above the Skin". JAMA Pediatr. 2016 Jan;170(1):9-10. doi: 10.1001/jamapediatrics.2015.2786. No abstract available. PMID 26595371
- [Background] Hill JO, Peters JC. Environmental contributions to the obesity epidemic. Science. 1998 May 29;280(5368):1371-4. doi: 10.1126/science.280.5368.1371. PMID 9603719
- [Background] Rodearmel SJ, Wyatt HR, Stroebele N, Smith SM, Ogden LG, Hill JO. Small changes in dietary sugar and physical activity as an approach to preventing excessive weight gain: the America on the Move family study. Pediatrics. 2007 Oct;120(4):e869-79. doi: 10.1542/peds.2006-2927. PMID 17908743
- [Background] Hill JO. Can a small-changes approach help address the obesity epidemic? A report of the Joint Task Force of the American Society for Nutrition, Institute of Food Technologists, and International Food Information Council. Am J Clin Nutr. 2009 Feb;89(2):477-84. doi: 10.3945/ajcn.2008.26566. Epub 2008 Dec 16. PMID 19088151
- [Background] Fisher JO, Birch LL. Restricting access to foods and children's eating. Appetite. 1999 Jun;32(3):405-19. doi: 10.1006/appe.1999.0231. PMID 10336797
- [Background] Hill C, Llewellyn CH, Saxton J, Webber L, Semmler C, Carnell S, van Jaarsveld CH, Boniface D, Wardle J. Adiposity and 'eating in the absence of hunger' in children. Int J Obes (Lond). 2008 Oct;32(10):1499-505. doi: 10.1038/ijo.2008.113. Epub 2008 Jul 22. PMID 18645573
- [Background] Fisher JO, Birch LL. Eating in the absence of hunger and overweight in girls from 5 to 7 y of age. Am J Clin Nutr. 2002 Jul;76(1):226-31. doi: 10.1093/ajcn/76.1.226. PMID 12081839
- [Background] Emond JA, Lansigan RK, Ramanujam A, Gilbert-Diamond D. Randomized Exposure to Food Advertisements and Eating in the Absence of Hunger Among Preschoolers. Pediatrics. 2016 Dec;138(6):e20162361. doi: 10.1542/peds.2016-2361. PMID 27940713
- [Background] Harris JL, Bargh JA, Brownell KD. Priming effects of television food advertising on eating behavior. Health Psychol. 2009 Jul;28(4):404-13. doi: 10.1037/a0014399. PMID 19594263
- [Background] Halford JC, Gillespie J, Brown V, Pontin EE, Dovey TM. Effect of television advertisements for foods on food consumption in children. Appetite. 2004 Apr;42(2):221-5. doi: 10.1016/j.appet.2003.11.006. PMID 15010186
- [Background] Halford JC, Boyland EJ, Hughes G, Oliveira LP, Dovey TM. Beyond-brand effect of television (TV) food advertisements/commercials on caloric intake and food choice of 5-7-year-old children. Appetite. 2007 Jul;49(1):263-7. doi: 10.1016/j.appet.2006.12.003. Epub 2006 Dec 23. PMID 17258351
- [Background] Halford JC, Boyland EJ, Hughes GM, Stacey L, McKean S, Dovey TM. Beyond-brand effect of television food advertisements on food choice in children: the effects of weight status. Public Health Nutr. 2008 Sep;11(9):897-904. doi: 10.1017/S1368980007001231. Epub 2007 Nov 16. PMID 18005487
- [Background] Anschutz DJ, Engels RC, Van Strien T. Side effects of television food commercials on concurrent nonadvertised sweet snack food intakes in young children. Am J Clin Nutr. 2009 May;89(5):1328-33. doi: 10.3945/ajcn.2008.27075. Epub 2009 Mar 25. PMID 19321557
- [Background] Bassareo V, Cucca F, Musio P, Lecca D, Frau R, Di Chiara G. Nucleus accumbens shell and core dopamine responsiveness to sucrose in rats: role of response contingency and discriminative/conditioned cues. Eur J Neurosci. 2015 Mar;41(6):802-9. doi: 10.1111/ejn.12839. Epub 2015 Feb 3. PMID 25645148
- [Background] Pavlov IP. Experimental Psychology and Psycho-Pathology in Animals. New York, New York: International Congress of Medicine; 1928. doi:10.1037/11081-001.
- [Background] Demos KE, Heatherton TF, Kelley WM. Individual differences in nucleus accumbens activity to food and sexual images predict weight gain and sexual behavior. J Neurosci. 2012 Apr 18;32(16):5549-52. doi: 10.1523/JNEUROSCI.5958-11.2012. PMID 22514316
- [Background] Volkow ND, Wang GJ, Fowler JS, Tomasi D. Addiction circuitry in the human brain. Annu Rev Pharmacol Toxicol. 2012;52:321-36. doi: 10.1146/annurev-pharmtox-010611-134625. Epub 2011 Sep 27. PMID 21961707
- [Background] Wagner DD, Boswell RG, Kelley WM, Heatherton TF. Inducing negative affect increases the reward value of appetizing foods in dieters. J Cogn Neurosci. 2012 Jul;24(7):1625-33. doi: 10.1162/jocn_a_00238. Epub 2012 Apr 23. PMID 22524295
- [Background] Stoeckel LE, Weller RE, Cook EW 3rd, Twieg DB, Knowlton RC, Cox JE. Widespread reward-system activation in obese women in response to pictures of high-calorie foods. Neuroimage. 2008 Jun;41(2):636-47. doi: 10.1016/j.neuroimage.2008.02.031. Epub 2008 Mar 4. PMID 18413289
- [Background] Castellanos EH, Charboneau E, Dietrich MS, Park S, Bradley BP, Mogg K, Cowan RL. Obese adults have visual attention bias for food cue images: evidence for altered reward system function. Int J Obes (Lond). 2009 Sep;33(9):1063-73. doi: 10.1038/ijo.2009.138. Epub 2009 Jul 21. PMID 19621020
- [Background] Lawrence NS, Hinton EC, Parkinson JA, Lawrence AD. Nucleus accumbens response to food cues predicts subsequent snack consumption in women and increased body mass index in those with reduced self-control. Neuroimage. 2012 Oct 15;63(1):415-22. doi: 10.1016/j.neuroimage.2012.06.070. Epub 2012 Jul 6. PMID 22776461
- [Background] Rapuano KM, Huckins JF, Sargent JD, Heatherton TF, Kelley WM. Individual Differences in Reward and Somatosensory-Motor Brain Regions Correlate with Adiposity in Adolescents. Cereb Cortex. 2016 Jun;26(6):2602-11. doi: 10.1093/cercor/bhv097. Epub 2015 May 20. PMID 25994961
- [Background] Rapuano KM, Zieselman AL, Kelley WM, Sargent JD, Heatherton TF, Gilbert-Diamond D. Genetic risk for obesity predicts nucleus accumbens size and responsivity to real-world food cues. Proc Natl Acad Sci U S A. 2017 Jan 3;114(1):160-165. doi: 10.1073/pnas.1605548113. Epub 2016 Dec 19. PMID 27994159
- [Background] Gearhardt AN, Yokum S, Stice E, Harris JL, Brownell KD. Relation of obesity to neural activation in response to food commercials. Soc Cogn Affect Neurosci. 2014 Jul;9(7):932-8. doi: 10.1093/scan/nst059. Epub 2013 Apr 10. PMID 23576811
- [Background] Stice E, Yokum S, Bohon C, Marti N, Smolen A. Reward circuitry responsivity to food predicts future increases in body mass: moderating effects of DRD2 and DRD4. Neuroimage. 2010 May 1;50(4):1618-25. doi: 10.1016/j.neuroimage.2010.01.081. Epub 2010 Jan 29. PMID 20116437
- [Background] Yokum S, Gearhardt AN, Harris JL, Brownell KD, Stice E. Individual differences in striatum activity to food commercials predict weight gain in adolescents. Obesity (Silver Spring). 2014 Dec;22(12):2544-51. doi: 10.1002/oby.20882. Epub 2014 Aug 25. PMID 25155745
- [Background] Zhao J, Bradfield JP, Li M, Wang K, Zhang H, Kim CE, Annaiah K, Glessner JT, Thomas K, Garris M, Frackelton EC, Otieno FG, Shaner JL, Smith RM, Chiavacci RM, Berkowitz RI, Hakonarson H, Grant SF. The role of obesity-associated loci identified in genome-wide association studies in the determination of pediatric BMI. Obesity (Silver Spring). 2009 Dec;17(12):2254-7. doi: 10.1038/oby.2009.159. Epub 2009 May 28. PMID 19478790
- [Background] den Hoed M, Ekelund U, Brage S, Grontved A, Zhao JH, Sharp SJ, Ong KK, Wareham NJ, Loos RJ. Genetic susceptibility to obesity and related traits in childhood and adolescence: influence of loci identified by genome-wide association studies. Diabetes. 2010 Nov;59(11):2980-8. doi: 10.2337/db10-0370. Epub 2010 Aug 19. PMID 20724581
- [Background] Willer CJ, Speliotes EK, Loos RJ, Li S, Lindgren CM, Heid IM, Berndt SI, Elliott AL, Jackson AU, Lamina C, Lettre G, Lim N, Lyon HN, McCarroll SA, Papadakis K, Qi L, Randall JC, Roccasecca RM, Sanna S, Scheet P, Weedon MN, Wheeler E, Zhao JH, Jacobs LC, Prokopenko I, Soranzo N, Tanaka T, Timpson NJ, Almgren P, Bennett A, Bergman RN, Bingham SA, Bonnycastle LL, Brown M, Burtt NP, Chines P, Coin L, Collins FS, Connell JM, Cooper C, Smith GD, Dennison EM, Deodhar P, Elliott P, Erdos MR, Estrada K, Evans DM, Gianniny L, Gieger C, Gillson CJ, Guiducci C, Hackett R, Hadley D, Hall AS, Havulinna AS, Hebebrand J, Hofman A, Isomaa B, Jacobs KB, Johnson T, Jousilahti P, Jovanovic Z, Khaw KT, Kraft P, Kuokkanen M, Kuusisto J, Laitinen J, Lakatta EG, Luan J, Luben RN, Mangino M, McArdle WL, Meitinger T, Mulas A, Munroe PB, Narisu N, Ness AR, Northstone K, O'Rahilly S, Purmann C, Rees MG, Ridderstrale M, Ring SM, Rivadeneira F, Ruokonen A, Sandhu MS, Saramies J, Scott LJ, Scuteri A, Silander K, Sims MA, Song K, Stephens J, Stevens S, Stringham HM, Tung YC, Valle TT, Van Duijn CM, Vimaleswaran KS, Vollenweider P, Waeber G, Wallace C, Watanabe RM, Waterworth DM, Watkins N; Wellcome Trust Case Control Consortium; Witteman JC, Zeggini E, Zhai G, Zillikens MC, Altshuler D, Caulfield MJ, Chanock SJ, Farooqi IS, Ferrucci L, Guralnik JM, Hattersley AT, Hu FB, Jarvelin MR, Laakso M, Mooser V, Ong KK, Ouwehand WH, Salomaa V, Samani NJ, Spector TD, Tuomi T, Tuomilehto J, Uda M, Uitterlinden AG, Wareham NJ, Deloukas P, Frayling TM, Groop LC, Hayes RB, Hunter DJ, Mohlke KL, Peltonen L, Schlessinger D, Strachan DP, Wichmann HE, McCarthy MI, Boehnke M, Barroso I, Abecasis GR, Hirschhorn JN; Genetic Investigation of ANthropometric Traits Consortium. Six new loci associated with body mass index highlight a neuronal influence on body weight regulation. Nat Genet. 2009 Jan;41(1):25-34. doi: 10.1038/ng.287. Epub 2008 Dec 14. PMID 19079261
- [Background] Thorleifsson G, Walters GB, Gudbjartsson DF, Steinthorsdottir V, Sulem P, Helgadottir A, Styrkarsdottir U, Gretarsdottir S, Thorlacius S, Jonsdottir I, Jonsdottir T, Olafsdottir EJ, Olafsdottir GH, Jonsson T, Jonsson F, Borch-Johnsen K, Hansen T, Andersen G, Jorgensen T, Lauritzen T, Aben KK, Verbeek AL, Roeleveld N, Kampman E, Yanek LR, Becker LC, Tryggvadottir L, Rafnar T, Becker DM, Gulcher J, Kiemeney LA, Pedersen O, Kong A, Thorsteinsdottir U, Stefansson K. Genome-wide association yields new sequence variants at seven loci that associate with measures of obesity. Nat Genet. 2009 Jan;41(1):18-24. doi: 10.1038/ng.274. Epub 2008 Dec 14. PMID 19079260
- [Background] Speliotes EK, Willer CJ, Berndt SI, Monda KL, Thorleifsson G, Jackson AU, Lango Allen H, Lindgren CM, Luan J, Magi R, Randall JC, Vedantam S, Winkler TW, Qi L, Workalemahu T, Heid IM, Steinthorsdottir V, Stringham HM, Weedon MN, Wheeler E, Wood AR, Ferreira T, Weyant RJ, Segre AV, Estrada K, Liang L, Nemesh J, Park JH, Gustafsson S, Kilpelainen TO, Yang J, Bouatia-Naji N, Esko T, Feitosa MF, Kutalik Z, Mangino M, Raychaudhuri S, Scherag A, Smith AV, Welch R, Zhao JH, Aben KK, Absher DM, Amin N, Dixon AL, Fisher E, Glazer NL, Goddard ME, Heard-Costa NL, Hoesel V, Hottenga JJ, Johansson A, Johnson T, Ketkar S, Lamina C, Li S, Moffatt MF, Myers RH, Narisu N, Perry JR, Peters MJ, Preuss M, Ripatti S, Rivadeneira F, Sandholt C, Scott LJ, Timpson NJ, Tyrer JP, van Wingerden S, Watanabe RM, White CC, Wiklund F, Barlassina C, Chasman DI, Cooper MN, Jansson JO, Lawrence RW, Pellikka N, Prokopenko I, Shi J, Thiering E, Alavere H, Alibrandi MT, Almgren P, Arnold AM, Aspelund T, Atwood LD, Balkau B, Balmforth AJ, Bennett AJ, Ben-Shlomo Y, Bergman RN, Bergmann S, Biebermann H, Blakemore AI, Boes T, Bonnycastle LL, Bornstein SR, Brown MJ, Buchanan TA, Busonero F, Campbell H, Cappuccio FP, Cavalcanti-Proenca C, Chen YD, Chen CM, Chines PS, Clarke R, Coin L, Connell J, Day IN, den Heijer M, Duan J, Ebrahim S, Elliott P, Elosua R, Eiriksdottir G, Erdos MR, Eriksson JG, Facheris MF, Felix SB, Fischer-Posovszky P, Folsom AR, Friedrich N, Freimer NB, Fu M, Gaget S, Gejman PV, Geus EJ, Gieger C, Gjesing AP, Goel A, Goyette P, Grallert H, Grassler J, Greenawalt DM, Groves CJ, Gudnason V, Guiducci C, Hartikainen AL, Hassanali N, Hall AS, Havulinna AS, Hayward C, Heath AC, Hengstenberg C, Hicks AA, Hinney A, Hofman A, Homuth G, Hui J, Igl W, Iribarren C, Isomaa B, Jacobs KB, Jarick I, Jewell E, John U, Jorgensen T, Jousilahti P, Jula A, Kaakinen M, Kajantie E, Kaplan LM, Kathiresan S, Kettunen J, Kinnunen L, Knowles JW, Kolcic I, Konig IR, Koskinen S, Kovacs P, Kuusisto J, Kraft P, Kvaloy K, Laitinen J, Lantieri O, Lanzani C, Launer LJ, Lecoeur C, Lehtimaki T, Lettre G, Liu J, Lokki ML, Lorentzon M, Luben RN, Ludwig B; MAGIC; Manunta P, Marek D, Marre M, Martin NG, McArdle WL, McCarthy A, McKnight B, Meitinger T, Melander O, Meyre D, Midthjell K, Montgomery GW, Morken MA, Morris AP, Mulic R, Ngwa JS, Nelis M, Neville MJ, Nyholt DR, O'Donnell CJ, O'Rahilly S, Ong KK, Oostra B, Pare G, Parker AN, Perola M, Pichler I, Pietilainen KH, Platou CG, Polasek O, Pouta A, Rafelt S, Raitakari O, Rayner NW, Ridderstrale M, Rief W, Ruokonen A, Robertson NR, Rzehak P, Salomaa V, Sanders AR, Sandhu MS, Sanna S, Saramies J, Savolainen MJ, Scherag S, Schipf S, Schreiber S, Schunkert H, Silander K, Sinisalo J, Siscovick DS, Smit JH, Soranzo N, Sovio U, Stephens J, Surakka I, Swift AJ, Tammesoo ML, Tardif JC, Teder-Laving M, Teslovich TM, Thompson JR, Thomson B, Tonjes A, Tuomi T, van Meurs JB, van Ommen GJ, Vatin V, Viikari J, Visvikis-Siest S, Vitart V, Vogel CI, Voight BF, Waite LL, Wallaschofski H, Walters GB, Widen E, Wiegand S, Wild SH, Willemsen G, Witte DR, Witteman JC, Xu J, Zhang Q, Zgaga L, Ziegler A, Zitting P, Beilby JP, Farooqi IS, Hebebrand J, Huikuri HV, James AL, Kahonen M, Levinson DF, Macciardi F, Nieminen MS, Ohlsson C, Palmer LJ, Ridker PM, Stumvoll M, Beckmann JS, Boeing H, Boerwinkle E, Boomsma DI, Caulfield MJ, Chanock SJ, Collins FS, Cupples LA, Smith GD, Erdmann J, Froguel P, Gronberg H, Gyllensten U, Hall P, Hansen T, Harris TB, Hattersley AT, Hayes RB, Heinrich J, Hu FB, Hveem K, Illig T, Jarvelin MR, Kaprio J, Karpe F, Khaw KT, Kiemeney LA, Krude H, Laakso M, Lawlor DA, Metspalu A, Munroe PB, Ouwehand WH, Pedersen O, Penninx BW, Peters A, Pramstaller PP, Quertermous T, Reinehr T, Rissanen A, Rudan I, Samani NJ, Schwarz PE, Shuldiner AR, Spector TD, Tuomilehto J, Uda M, Uitterlinden A, Valle TT, Wabitsch M, Waeber G, Wareham NJ, Watkins H; Procardis Consortium; Wilson JF, Wright AF, Zillikens MC, Chatterjee N, McCarroll SA, Purcell S, Schadt EE, Visscher PM, Assimes TL, Borecki IB, Deloukas P, Fox CS, Groop LC, Haritunians T, Hunter DJ, Kaplan RC, Mohlke KL, O'Connell JR, Peltonen L, Schlessinger D, Strachan DP, van Duijn CM, Wichmann HE, Frayling TM, Thorsteinsdottir U, Abecasis GR, Barroso I, Boehnke M, Stefansson K, North KE, McCarthy MI, Hirschhorn JN, Ingelsson E, Loos RJ. Association analyses of 249,796 individuals reveal 18 new loci associated with body mass index. Nat Genet. 2010 Nov;42(11):937-48. doi: 10.1038/ng.686. Epub 2010 Oct 10. PMID 20935630
- [Background] Locke AE, Kahali B, Berndt SI, Justice AE, Pers TH, Day FR, Powell C, Vedantam S, Buchkovich ML, Yang J, Croteau-Chonka DC, Esko T, Fall T, Ferreira T, Gustafsson S, Kutalik Z, Luan J, Magi R, Randall JC, Winkler TW, Wood AR, Workalemahu T, Faul JD, Smith JA, Zhao JH, Zhao W, Chen J, Fehrmann R, Hedman AK, Karjalainen J, Schmidt EM, Absher D, Amin N, Anderson D, Beekman M, Bolton JL, Bragg-Gresham JL, Buyske S, Demirkan A, Deng G, Ehret GB, Feenstra B, Feitosa MF, Fischer K, Goel A, Gong J, Jackson AU, Kanoni S, Kleber ME, Kristiansson K, Lim U, Lotay V, Mangino M, Leach IM, Medina-Gomez C, Medland SE, Nalls MA, Palmer CD, Pasko D, Pechlivanis S, Peters MJ, Prokopenko I, Shungin D, Stancakova A, Strawbridge RJ, Sung YJ, Tanaka T, Teumer A, Trompet S, van der Laan SW, van Setten J, Van Vliet-Ostaptchouk JV, Wang Z, Yengo L, Zhang W, Isaacs A, Albrecht E, Arnlov J, Arscott GM, Attwood AP, Bandinelli S, Barrett A, Bas IN, Bellis C, Bennett AJ, Berne C, Blagieva R, Bluher M, Bohringer S, Bonnycastle LL, Bottcher Y, Boyd HA, Bruinenberg M, Caspersen IH, Chen YI, Clarke R, Daw EW, de Craen AJM, Delgado G, Dimitriou M, Doney ASF, Eklund N, Estrada K, Eury E, Folkersen L, Fraser RM, Garcia ME, Geller F, Giedraitis V, Gigante B, Go AS, Golay A, Goodall AH, Gordon SD, Gorski M, Grabe HJ, Grallert H, Grammer TB, Grassler J, Gronberg H, Groves CJ, Gusto G, Haessler J, Hall P, Haller T, Hallmans G, Hartman CA, Hassinen M, Hayward C, Heard-Costa NL, Helmer Q, Hengstenberg C, Holmen O, Hottenga JJ, James AL, Jeff JM, Johansson A, Jolley J, Juliusdottir T, Kinnunen L, Koenig W, Koskenvuo M, Kratzer W, Laitinen J, Lamina C, Leander K, Lee NR, Lichtner P, Lind L, Lindstrom J, Lo KS, Lobbens S, Lorbeer R, Lu Y, Mach F, Magnusson PKE, Mahajan A, McArdle WL, McLachlan S, Menni C, Merger S, Mihailov E, Milani L, Moayyeri A, Monda KL, Morken MA, Mulas A, Muller G, Muller-Nurasyid M, Musk AW, Nagaraja R, Nothen MM, Nolte IM, Pilz S, Rayner NW, Renstrom F, Rettig R, Ried JS, Ripke S, Robertson NR, Rose LM, Sanna S, Scharnagl H, Scholtens S, Schumacher FR, Scott WR, Seufferlein T, Shi J, Smith AV, Smolonska J, Stanton AV, Steinthorsdottir V, Stirrups K, Stringham HM, Sundstrom J, Swertz MA, Swift AJ, Syvanen AC, Tan ST, Tayo BO, Thorand B, Thorleifsson G, Tyrer JP, Uh HW, Vandenput L, Verhulst FC, Vermeulen SH, Verweij N, Vonk JM, Waite LL, Warren HR, Waterworth D, Weedon MN, Wilkens LR, Willenborg C, Wilsgaard T, Wojczynski MK, Wong A, Wright AF, Zhang Q; LifeLines Cohort Study; Brennan EP, Choi M, Dastani Z, Drong AW, Eriksson P, Franco-Cereceda A, Gadin JR, Gharavi AG, Goddard ME, Handsaker RE, Huang J, Karpe F, Kathiresan S, Keildson S, Kiryluk K, Kubo M, Lee JY, Liang L, Lifton RP, Ma B, McCarroll SA, McKnight AJ, Min JL, Moffatt MF, Montgomery GW, Murabito JM, Nicholson G, Nyholt DR, Okada Y, Perry JRB, Dorajoo R, Reinmaa E, Salem RM, Sandholm N, Scott RA, Stolk L, Takahashi A, Tanaka T, van 't Hooft FM, Vinkhuyzen AAE, Westra HJ, Zheng W, Zondervan KT; ADIPOGen Consortium; AGEN-BMI Working Group; CARDIOGRAMplusC4D Consortium; CKDGen Consortium; GLGC; ICBP; MAGIC Investigators; MuTHER Consortium; MIGen Consortium; PAGE Consortium; ReproGen Consortium; GENIE Consortium; International Endogene Consortium; Heath AC, Arveiler D, Bakker SJL, Beilby J, Bergman RN, Blangero J, Bovet P, Campbell H, Caulfield MJ, Cesana G, Chakravarti A, Chasman DI, Chines PS, Collins FS, Crawford DC, Cupples LA, Cusi D, Danesh J, de Faire U, den Ruijter HM, Dominiczak AF, Erbel R, Erdmann J, Eriksson JG, Farrall M, Felix SB, Ferrannini E, Ferrieres J, Ford I, Forouhi NG, Forrester T, Franco OH, Gansevoort RT, Gejman PV, Gieger C, Gottesman O, Gudnason V, Gyllensten U, Hall AS, Harris TB, Hattersley AT, Hicks AA, Hindorff LA, Hingorani AD, Hofman A, Homuth G, Hovingh GK, Humphries SE, Hunt SC, Hypponen E, Illig T, Jacobs KB, Jarvelin MR, Jockel KH, Johansen B, Jousilahti P, Jukema JW, Jula AM, Kaprio J, Kastelein JJP, Keinanen-Kiukaanniemi SM, Kiemeney LA, Knekt P, Kooner JS, Kooperberg C, Kovacs P, Kraja AT, Kumari M, Kuusisto J, Lakka TA, Langenberg C, Marchand LL, Lehtimaki T, Lyssenko V, Mannisto S, Marette A, Matise TC, McKenzie CA, McKnight B, Moll FL, Morris AD, Morris AP, Murray JC, Nelis M, Ohlsson C, Oldehinkel AJ, Ong KK, Madden PAF, Pasterkamp G, Peden JF, Peters A, Postma DS, Pramstaller PP, Price JF, Qi L, Raitakari OT, Rankinen T, Rao DC, Rice TK, Ridker PM, Rioux JD, Ritchie MD, Rudan I, Salomaa V, Samani NJ, Saramies J, Sarzynski MA, Schunkert H, Schwarz PEH, Sever P, Shuldiner AR, Sinisalo J, Stolk RP, Strauch K, Tonjes A, Tregouet DA, Tremblay A, Tremoli E, Virtamo J, Vohl MC, Volker U, Waeber G, Willemsen G, Witteman JC, Zillikens MC, Adair LS, Amouyel P, Asselbergs FW, Assimes TL, Bochud M, Boehm BO, Boerwinkle E, Bornstein SR, Bottinger EP, Bouchard C, Cauchi S, Chambers JC, Chanock SJ, Cooper RS, de Bakker PIW, Dedoussis G, Ferrucci L, Franks PW, Froguel P, Groop LC, Haiman CA, Hamsten A, Hui J, Hunter DJ, Hveem K, Kaplan RC, Kivimaki M, Kuh D, Laakso M, Liu Y, Martin NG, Marz W, Melbye M, Metspalu A, Moebus S, Munroe PB, Njolstad I, Oostra BA, Palmer CNA, Pedersen NL, Perola M, Perusse L, Peters U, Power C, Quertermous T, Rauramaa R, Rivadeneira F, Saaristo TE, Saleheen D, Sattar N, Schadt EE, Schlessinger D, Slagboom PE, Snieder H, Spector TD, Thorsteinsdottir U, Stumvoll M, Tuomilehto J, Uitterlinden AG, Uusitupa M, van der Harst P, Walker M, Wallaschofski H, Wareham NJ, Watkins H, Weir DR, Wichmann HE, Wilson JF, Zanen P, Borecki IB, Deloukas P, Fox CS, Heid IM, O'Connell JR, Strachan DP, Stefansson K, van Duijn CM, Abecasis GR, Franke L, Frayling TM, McCarthy MI, Visscher PM, Scherag A, Willer CJ, Boehnke M, Mohlke KL, Lindgren CM, Beckmann JS, Barroso I, North KE, Ingelsson E, Hirschhorn JN, Loos RJF, Speliotes EK. Genetic studies of body mass index yield new insights for obesity biology. Nature. 2015 Feb 12;518(7538):197-206. doi: 10.1038/nature14177. PMID 25673413
- [Background] Hess ME, Hess S, Meyer KD, Verhagen LA, Koch L, Bronneke HS, Dietrich MO, Jordan SD, Saletore Y, Elemento O, Belgardt BF, Franz T, Horvath TL, Ruther U, Jaffrey SR, Kloppenburg P, Bruning JC. The fat mass and obesity associated gene (Fto) regulates activity of the dopaminergic midbrain circuitry. Nat Neurosci. 2013 Aug;16(8):1042-8. doi: 10.1038/nn.3449. Epub 2013 Jun 30. PMID 23817550
- [Background] Wardle J, Llewellyn C, Sanderson S, Plomin R. The FTO gene and measured food intake in children. Int J Obes (Lond). 2009 Jan;33(1):42-5. doi: 10.1038/ijo.2008.174. Epub 2008 Oct 7. PMID 18838977
- [Background] Carnell S, Wardle J. Appetite and adiposity in children: evidence for a behavioral susceptibility theory of obesity. Am J Clin Nutr. 2008 Jul;88(1):22-9. doi: 10.1093/ajcn/88.1.22. PMID 18614720
- [Background] Wardle J, Carnell S, Haworth CM, Farooqi IS, O'Rahilly S, Plomin R. Obesity associated genetic variation in FTO is associated with diminished satiety. J Clin Endocrinol Metab. 2008 Sep;93(9):3640-3. doi: 10.1210/jc.2008-0472. Epub 2008 Jun 26. PMID 18583465
- [Background] Smemo S, Tena JJ, Kim KH, Gamazon ER, Sakabe NJ, Gomez-Marin C, Aneas I, Credidio FL, Sobreira DR, Wasserman NF, Lee JH, Puviindran V, Tam D, Shen M, Son JE, Vakili NA, Sung HK, Naranjo S, Acemel RD, Manzanares M, Nagy A, Cox NJ, Hui CC, Gomez-Skarmeta JL, Nobrega MA. Obesity-associated variants within FTO form long-range functional connections with IRX3. Nature. 2014 Mar 20;507(7492):371-5. doi: 10.1038/nature13138. Epub 2014 Mar 12. PMID 24646999
- [Background] Ho-Urriola J, Guzman-Guzman IP, Smalley SV, Gonzalez A, Weisstaub G, Dominguez-Vasquez P, Valladares M, Amador P, Hodgson MI, Obregon AM, Santos JL. Melanocortin-4 receptor polymorphism rs17782313: association with obesity and eating in the absence of hunger in Chilean children. Nutrition. 2014 Feb;30(2):145-9. doi: 10.1016/j.nut.2013.05.030. Epub 2013 Oct 15. PMID 24139164
- [Background] Llewellyn CH, Trzaskowski M, van Jaarsveld CHM, Plomin R, Wardle J. Satiety mechanisms in genetic risk of obesity. JAMA Pediatr. 2014 Apr;168(4):338-344. doi: 10.1001/jamapediatrics.2013.4944. PMID 24535189
- [Background] Elks CE, Loos RJ, Sharp SJ, Langenberg C, Ring SM, Timpson NJ, Ness AR, Davey Smith G, Dunger DB, Wareham NJ, Ong KK. Genetic markers of adult obesity risk are associated with greater early infancy weight gain and growth. PLoS Med. 2010 May 25;7(5):e1000284. doi: 10.1371/journal.pmed.1000284. PMID 20520848
- [Background] Belsky DW, Moffitt TE, Houts R, Bennett GG, Biddle AK, Blumenthal JA, Evans JP, Harrington H, Sugden K, Williams B, Poulton R, Caspi A. Polygenic risk, rapid childhood growth, and the development of obesity: evidence from a 4-decade longitudinal study. Arch Pediatr Adolesc Med. 2012 Jun 1;166(6):515-21. doi: 10.1001/archpediatrics.2012.131. PMID 22665028
- [Background] Elks CE, Loos RJ, Hardy R, Wills AK, Wong A, Wareham NJ, Kuh D, Ong KK. Adult obesity susceptibility variants are associated with greater childhood weight gain and a faster tempo of growth: the 1946 British Birth Cohort Study. Am J Clin Nutr. 2012 May;95(5):1150-6. doi: 10.3945/ajcn.111.027870. Epub 2012 Mar 28. PMID 22456663
- [Background] Field AE, Camargo CA Jr, Ogino S. The merits of subtyping obesity: one size does not fit all. JAMA. 2013 Nov 27;310(20):2147-8. doi: 10.1001/jama.2013.281501. No abstract available. PMID 24189835
- [Background] Seeyave DM, Coleman S, Appugliese D, Corwyn RF, Bradley RH, Davidson NS, Kaciroti N, Lumeng JC. Ability to delay gratification at age 4 years and risk of overweight at age 11 years. Arch Pediatr Adolesc Med. 2009 Apr;163(4):303-8. doi: 10.1001/archpediatrics.2009.12. PMID 19349558
- [Background] Francis LA, Susman EJ. Self-regulation and rapid weight gain in children from age 3 to 12 years. Arch Pediatr Adolesc Med. 2009 Apr;163(4):297-302. doi: 10.1001/archpediatrics.2008.579. PMID 19349557
- [Background] Duckworth AL, Tsukayama E, Geier AB. Self-controlled children stay leaner in the transition to adolescence. Appetite. 2010 Apr;54(2):304-8. doi: 10.1016/j.appet.2009.11.016. Epub 2009 Dec 11. PMID 20004223
- [Background] Tsukayama E, Toomey SL, Faith MS, Duckworth AL. Self-control as a protective factor against overweight status in the transition from childhood to adolescence. Arch Pediatr Adolesc Med. 2010 Jul;164(7):631-5. doi: 10.1001/archpediatrics.2010.97. PMID 20603463
- [Background] Grolnick WS, Ryan RM. Parent styles associated with children's self-regulation and competence in school. Journal of Educational Psychology. 1989;81(2):143-154. doi:10.1037/0022-0663.81.2.143.
- [Background] Dahlgren CL, Lask B, Landro NI, Ro O. Patient and parental self-reports of executive functioning in a sample of young female adolescents with anorexia nervosa before and after cognitive remediation therapy. Eur Eat Disord Rev. 2014 Jan;22(1):45-52. doi: 10.1002/erv.2265. Epub 2013 Oct 16. PMID 24129969
- [Background] Anzman SL, Birch LL. Low inhibitory control and restrictive feeding practices predict weight outcomes. J Pediatr. 2009 Nov;155(5):651-6. doi: 10.1016/j.jpeds.2009.04.052. PMID 19595373
- [Background] Duckworth AL, Seligman ME. Self-discipline outdoes IQ in predicting academic performance of adolescents. Psychol Sci. 2005 Dec;16(12):939-44. doi: 10.1111/j.1467-9280.2005.01641.x. PMID 16313657
- [Background] Best JR, Miller PH. A developmental perspective on executive function. Child Dev. 2010 Nov-Dec;81(6):1641-60. doi: 10.1111/j.1467-8624.2010.01499.x. PMID 21077853
- [Background] Hassin RR, Ochsner KNKN, Trope Y. The common neural basis for exerting self-control in different domains. In: Oxford ; New York : Oxford University Press; 2010:141-162.
- [Background] Stang J, Loth KA. Parenting style and child feeding practices: potential mitigating factors in the etiology of childhood obesity. J Am Diet Assoc. 2011 Sep;111(9):1301-5. doi: 10.1016/j.jada.2011.06.010. No abstract available. PMID 21872692
- [Background] Rollins BY, Savage JS, Fisher JO, Birch LL. Alternatives to restrictive feeding practices to promote self-regulation in childhood: a developmental perspective. Pediatr Obes. 2016 Oct;11(5):326-32. doi: 10.1111/ijpo.12071. Epub 2015 Sep 25. PMID 26403816
- [Background] Rodgers RF, Paxton SJ, Massey R, Campbell KJ, Wertheim EH, Skouteris H, Gibbons K. Maternal feeding practices predict weight gain and obesogenic eating behaviors in young children: a prospective study. Int J Behav Nutr Phys Act. 2013 Feb 18;10:24. doi: 10.1186/1479-5868-10-24. PMID 23414332
- [Background] Faith MS, Scanlon KS, Birch LL, Francis LA, Sherry B. Parent-child feeding strategies and their relationships to child eating and weight status. Obes Res. 2004 Nov;12(11):1711-22. doi: 10.1038/oby.2004.212. PMID 15601964
- [Background] Gubbels JS, Kremers SP, Stafleu A, de Vries SI, Goldbohm RA, Dagnelie PC, de Vries NK, van Buuren S, Thijs C. Association between parenting practices and children's dietary intake, activity behavior and development of body mass index: the KOALA Birth Cohort Study. Int J Behav Nutr Phys Act. 2011 Mar 14;8:18. doi: 10.1186/1479-5868-8-18. PMID 21401954
- [Background] Rollins BY, Loken E, Savage JS, Birch LL. Measurement of food reinforcement in preschool children. Associations with food intake, BMI, and reward sensitivity. Appetite. 2014 Jan;72:21-7. doi: 10.1016/j.appet.2013.09.018. Epub 2013 Sep 30. PMID 24090537
- [Background] Powers SW, Chamberlin LA, van Schaick KB, Sherman SN, Whitaker RC. Maternal feeding strategies, child eating behaviors, and child BMI in low-income African-American preschoolers. Obesity (Silver Spring). 2006 Nov;14(11):2026-33. doi: 10.1038/oby.2006.237. PMID 17135620
- [Background] Tovar A, Emond JA, Hennessy E, Gilbert-Diamond D. An FTO Gene Variant Moderates the Association between Parental Restriction and Child BMI. PLoS One. 2016 May 19;11(5):e0155521. doi: 10.1371/journal.pone.0155521. eCollection 2016. PMID 27196523
- [Background] Allen HA, Chambers A, Blissett J, Chechlacz M, Barrett T, Higgs S, Nouwen A. Relationship between Parental Feeding Practices and Neural Responses to Food Cues in Adolescents. PLoS One. 2016 Aug 1;11(8):e0157037. doi: 10.1371/journal.pone.0157037. eCollection 2016. PMID 27479051
- [Background] Shloim N, Edelson LR, Martin N, Hetherington MM. Parenting Styles, Feeding Styles, Feeding Practices, and Weight Status in 4-12 Year-Old Children: A Systematic Review of the Literature. Front Psychol. 2015 Dec 14;6:1849. doi: 10.3389/fpsyg.2015.01849. eCollection 2015. PMID 26696920
- [Background] Rideout VJ. The Common Sense Census: Media Use by Tweens and Teens. Common Sense Media. https://www.commonsensemedia.org/sites/default/files/uploads/research/census_executivesummary.pdf. Published October 21, 2015. Accessed July 5, 2017.
- [Background] Frazier WC, Harris JL. Trends in Television Food Advertising to Young People: 2016 Update. UConn Rudd Center for Food Policy and Obesity. http://www.uconnruddcenter.org/files/TVAdTrends2017.pdf. Published June 2017. Accessed June 15, 2017.
- [Background] Botha S, Fentonmiller K, Jennings C, Johnson M, Rusk MK, Young K. A Review of Food Marketing to Children and Adolescents: Follow-Up Report. Washington, DC: Federal Trade Commission; 2012.
- [Background] Rideout VJ. Advertising to Children and Teens: Current Practices. Common Sense Media.
- [Background] Ustjanauskas AE, Harris JL, Schwartz MB. Food and beverage advertising on children's web sites. Pediatr Obes. 2014 Oct;9(5):362-72. doi: 10.1111/j.2047-6310.2013.00185.x. Epub 2013 Jul 2. PMID 23818245
- [Background] National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. Preventing Tobacco Use Among Youth and Young Adults: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK99237/ PMID 22876391
- [Background] Sargent JD, Heatherton TF. Comparison of trends for adolescent smoking and smoking in movies, 1990-2007. JAMA. 2009 Jun 3;301(21):2211-3. doi: 10.1001/jama.2009.745. No abstract available. PMID 19491181
- [Background] Heatherton TF, Sargent JD. Does Watching Smoking in Movies Promote Teenage Smoking? Curr Dir Psychol Sci. 2009 Apr 15;18(2):63-67. doi: 10.1111/j.1467-8721.2009.01610.x. PMID 20160916
- [Background] Wiemerslage L, Nilsson EK, Solstrand Dahlberg L, Ence-Eriksson F, Castillo S, Larsen AL, Bylund SB, Hogenkamp PS, Olivo G, Bandstein M, Titova OE, Larsson EM, Benedict C, Brooks SJ, Schioth HB. An obesity-associated risk allele within the FTO gene affects human brain activity for areas important for emotion, impulse control and reward in response to food images. Eur J Neurosci. 2016 May;43(9):1173-80. doi: 10.1111/ejn.13177. Epub 2016 Feb 21. PMID 26797854
- [Background] van der Klaauw AA, von dem Hagen EA, Keogh JM, Henning E, O'Rahilly S, Lawrence AD, Calder AJ, Farooqi IS. Obesity-associated melanocortin-4 receptor mutations are associated with changes in the brain response to food cues. J Clin Endocrinol Metab. 2014 Oct;99(10):E2101-6. doi: 10.1210/jc.2014-1651. Epub 2014 Jul 25. PMID 25062455
- [Background] Baicy K, London ED, Monterosso J, Wong ML, Delibasi T, Sharma A, Licinio J. Leptin replacement alters brain response to food cues in genetically leptin-deficient adults. Proc Natl Acad Sci U S A. 2007 Nov 13;104(46):18276-9. doi: 10.1073/pnas.0706481104. Epub 2007 Nov 6. PMID 17986612
- [Background] Kuhn AB, Feis DL, Schilbach L, Kracht L, Hess ME, Mauer J, Bruning JC, Tittgemeyer M. FTO gene variant modulates the neural correlates of visual food perception. Neuroimage. 2016 Mar;128:21-31. doi: 10.1016/j.neuroimage.2015.12.049. Epub 2016 Jan 5. PMID 26767945
- [Background] Gilbert-Diamond D, Moore JH. Analysis of Gene-Gene Interactions. Hoboken, NJ, USA: John Wiley & Sons, Inc.; 2011:1.14.1-1.14.12. doi:10.1002/0471142905.hg0114s70.
- [Background] Centers for Disease Control and Prevention. CDC Growth Charts: United States. Washington, DC; 2000. http://www.cdc.gov/growthcharts/.
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- [Background] Birch LL, Fisher JO, Grimm-Thomas K, Markey CN, Sawyer R, Johnson SL. Confirmatory factor analysis of the Child Feeding Questionnaire: a measure of parental attitudes, beliefs and practices about child feeding and obesity proneness. Appetite. 2001 Jun;36(3):201-10. doi: 10.1006/appe.2001.0398. PMID 11358344
- [Background] Frayling TM, Timpson NJ, Weedon MN, Zeggini E, Freathy RM, Lindgren CM, Perry JR, Elliott KS, Lango H, Rayner NW, Shields B, Harries LW, Barrett JC, Ellard S, Groves CJ, Knight B, Patch AM, Ness AR, Ebrahim S, Lawlor DA, Ring SM, Ben-Shlomo Y, Jarvelin MR, Sovio U, Bennett AJ, Melzer D, Ferrucci L, Loos RJ, Barroso I, Wareham NJ, Karpe F, Owen KR, Cardon LR, Walker M, Hitman GA, Palmer CN, Doney AS, Morris AD, Smith GD, Hattersley AT, McCarthy MI. A common variant in the FTO gene is associated with body mass index and predisposes to childhood and adult obesity. Science. 2007 May 11;316(5826):889-94. doi: 10.1126/science.1141634. Epub 2007 Apr 12. PMID 17434869
- [Background] Benjamini Y, Hochberg Y. Controlling the false discovery rate: a practical and powerful approach to multiple testing. Journal of the royal statistical society Series B. 1995. doi:10.2307/2346101.
- [Background] Bernhardt AM, Wilking C, Gottlieb M, Emond J, Sargent JD. Children's reaction to depictions of healthy foods in fast-food television advertisements. JAMA Pediatr. 2014 May;168(5):422-6. doi: 10.1001/jamapediatrics.2014.140. PMID 24686476
- [Background] Illumina. Infinium Global Screening Array-24 v1.0 BeadChip. https://www.illumina.com/content/dam/illumina-marketing/documents/products/datasheets/infinium-commercial-gsa-data-sheet-370-2016-016.pdf. Published March 29, 2017. Accessed June 1, 2017.
- [Background] Graff M, Scott RA, Justice AE, Young KL, Feitosa MF, Barata L, Winkler TW, Chu AY, Mahajan A, Hadley D, Xue L, Workalemahu T, Heard-Costa NL, den Hoed M, Ahluwalia TS, Qi Q, Ngwa JS, Renstrom F, Quaye L, Eicher JD, Hayes JE, Cornelis M, Kutalik Z, Lim E, Luan J, Huffman JE, Zhang W, Zhao W, Griffin PJ, Haller T, Ahmad S, Marques-Vidal PM, Bien S, Yengo L, Teumer A, Smith AV, Kumari M, Harder MN, Justesen JM, Kleber ME, Hollensted M, Lohman K, Rivera NV, Whitfield JB, Zhao JH, Stringham HM, Lyytikainen LP, Huppertz C, Willemsen G, Peyrot WJ, Wu Y, Kristiansson K, Demirkan A, Fornage M, Hassinen M, Bielak LF, Cadby G, Tanaka T, Magi R, van der Most PJ, Jackson AU, Bragg-Gresham JL, Vitart V, Marten J, Navarro P, Bellis C, Pasko D, Johansson A, Snitker S, Cheng YC, Eriksson J, Lim U, Aadahl M, Adair LS, Amin N, Balkau B, Auvinen J, Beilby J, Bergman RN, Bergmann S, Bertoni AG, Blangero J, Bonnefond A, Bonnycastle LL, Borja JB, Brage S, Busonero F, Buyske S, Campbell H, Chines PS, Collins FS, Corre T, Smith GD, Delgado GE, Dueker N, Dorr M, Ebeling T, Eiriksdottir G, Esko T, Faul JD, Fu M, Faerch K, Gieger C, Glaser S, Gong J, Gordon-Larsen P, Grallert H, Grammer TB, Grarup N, van Grootheest G, Harald K, Hastie ND, Havulinna AS, Hernandez D, Hindorff L, Hocking LJ, Holmens OL, Holzapfel C, Hottenga JJ, Huang J, Huang T, Hui J, Huth C, Hutri-Kahonen N, James AL, Jansson JO, Jhun MA, Juonala M, Kinnunen L, Koistinen HA, Kolcic I, Komulainen P, Kuusisto J, Kvaloy K, Kahonen M, Lakka TA, Launer LJ, Lehne B, Lindgren CM, Lorentzon M, Luben R, Marre M, Milaneschi Y, Monda KL, Montgomery GW, De Moor MHM, Mulas A, Muller-Nurasyid M, Musk AW, Mannikko R, Mannisto S, Narisu N, Nauck M, Nettleton JA, Nolte IM, Oldehinkel AJ, Olden M, Ong KK, Padmanabhan S, Paternoster L, Perez J, Perola M, Peters A, Peters U, Peyser PA, Prokopenko I, Puolijoki H, Raitakari OT, Rankinen T, Rasmussen-Torvik LJ, Rawal R, Ridker PM, Rose LM, Rudan I, Sarti C, Sarzynski MA, Savonen K, Scott WR, Sanna S, Shuldiner AR, Sidney S, Silbernagel G, Smith BH, Smith JA, Snieder H, Stancakova A, Sternfeld B, Swift AJ, Tammelin T, Tan ST, Thorand B, Thuillier D, Vandenput L, Vestergaard H, van Vliet-Ostaptchouk JV, Vohl MC, Volker U, Waeber G, Walker M, Wild S, Wong A, Wright AF, Zillikens MC, Zubair N, Haiman CA, Lemarchand L, Gyllensten U, Ohlsson C, Hofman A, Rivadeneira F, Uitterlinden AG, Perusse L, Wilson JF, Hayward C, Polasek O, Cucca F, Hveem K, Hartman CA, Tonjes A, Bandinelli S, Palmer LJ, Kardia SLR, Rauramaa R, Sorensen TIA, Tuomilehto J, Salomaa V, Penninx BWJH, de Geus EJC, Boomsma DI, Lehtimaki T, Mangino M, Laakso M, Bouchard C, Martin NG, Kuh D, Liu Y, Linneberg A, Marz W, Strauch K, Kivimaki M, Harris TB, Gudnason V, Volzke H, Qi L, Jarvelin MR, Chambers JC, Kooner JS, Froguel P, Kooperberg C, Vollenweider P, Hallmans G, Hansen T, Pedersen O, Metspalu A, Wareham NJ, Langenberg C, Weir DR, Porteous DJ, Boerwinkle E, Chasman DI; CHARGE Consortium; EPIC-InterAct Consortium; PAGE Consortium; Abecasis GR, Barroso I, McCarthy MI, Frayling TM, O'Connell JR, van Duijn CM, Boehnke M, Heid IM, Mohlke KL, Strachan DP, Fox CS, Liu CT, Hirschhorn JN, Klein RJ, Johnson AD, Borecki IB, Franks PW, North KE, Cupples LA, Loos RJF, Kilpelainen TO. Genome-wide physical activity interactions in adiposity - A meta-analysis of 200,452 adults. PLoS Genet. 2017 Apr 27;13(4):e1006528. doi: 10.1371/journal.pgen.1006528. eCollection 2017 Apr. PMID 28448500
- [Background] Justice AE, Winkler TW, Feitosa MF, Graff M, Fisher VA, Young K, Barata L, Deng X, Czajkowski J, Hadley D, Ngwa JS, Ahluwalia TS, Chu AY, Heard-Costa NL, Lim E, Perez J, Eicher JD, Kutalik Z, Xue L, Mahajan A, Renstrom F, Wu J, Qi Q, Ahmad S, Alfred T, Amin N, Bielak LF, Bonnefond A, Bragg J, Cadby G, Chittani M, Coggeshall S, Corre T, Direk N, Eriksson J, Fischer K, Gorski M, Neergaard Harder M, Horikoshi M, Huang T, Huffman JE, Jackson AU, Justesen JM, Kanoni S, Kinnunen L, Kleber ME, Komulainen P, Kumari M, Lim U, Luan J, Lyytikainen LP, Mangino M, Manichaikul A, Marten J, Middelberg RPS, Muller-Nurasyid M, Navarro P, Perusse L, Pervjakova N, Sarti C, Smith AV, Smith JA, Stancakova A, Strawbridge RJ, Stringham HM, Sung YJ, Tanaka T, Teumer A, Trompet S, van der Laan SW, van der Most PJ, Van Vliet-Ostaptchouk JV, Vedantam SL, Verweij N, Vink JM, Vitart V, Wu Y, Yengo L, Zhang W, Hua Zhao J, Zimmermann ME, Zubair N, Abecasis GR, Adair LS, Afaq S, Afzal U, Bakker SJL, Bartz TM, Beilby J, Bergman RN, Bergmann S, Biffar R, Blangero J, Boerwinkle E, Bonnycastle LL, Bottinger E, Braga D, Buckley BM, Buyske S, Campbell H, Chambers JC, Collins FS, Curran JE, de Borst GJ, de Craen AJM, de Geus EJC, Dedoussis G, Delgado GE, den Ruijter HM, Eiriksdottir G, Eriksson AL, Esko T, Faul JD, Ford I, Forrester T, Gertow K, Gigante B, Glorioso N, Gong J, Grallert H, Grammer TB, Grarup N, Haitjema S, Hallmans G, Hamsten A, Hansen T, Harris TB, Hartman CA, Hassinen M, Hastie ND, Heath AC, Hernandez D, Hindorff L, Hocking LJ, Hollensted M, Holmen OL, Homuth G, Jan Hottenga J, Huang J, Hung J, Hutri-Kahonen N, Ingelsson E, James AL, Jansson JO, Jarvelin MR, Jhun MA, Jorgensen ME, Juonala M, Kahonen M, Karlsson M, Koistinen HA, Kolcic I, Kolovou G, Kooperberg C, Kramer BK, Kuusisto J, Kvaloy K, Lakka TA, Langenberg C, Launer LJ, Leander K, Lee NR, Lind L, Lindgren CM, Linneberg A, Lobbens S, Loh M, Lorentzon M, Luben R, Lubke G, Ludolph-Donislawski A, Lupoli S, Madden PAF, Mannikko R, Marques-Vidal P, Martin NG, McKenzie CA, McKnight B, Mellstrom D, Menni C, Montgomery GW, Musk AB, Narisu N, Nauck M, Nolte IM, Oldehinkel AJ, Olden M, Ong KK, Padmanabhan S, Peyser PA, Pisinger C, Porteous DJ, Raitakari OT, Rankinen T, Rao DC, Rasmussen-Torvik LJ, Rawal R, Rice T, Ridker PM, Rose LM, Bien SA, Rudan I, Sanna S, Sarzynski MA, Sattar N, Savonen K, Schlessinger D, Scholtens S, Schurmann C, Scott RA, Sennblad B, Siemelink MA, Silbernagel G, Slagboom PE, Snieder H, Staessen JA, Stott DJ, Swertz MA, Swift AJ, Taylor KD, Tayo BO, Thorand B, Thuillier D, Tuomilehto J, Uitterlinden AG, Vandenput L, Vohl MC, Volzke H, Vonk JM, Waeber G, Waldenberger M, Westendorp RGJ, Wild S, Willemsen G, Wolffenbuttel BHR, Wong A, Wright AF, Zhao W, Zillikens MC, Baldassarre D, Balkau B, Bandinelli S, Boger CA, Boomsma DI, Bouchard C, Bruinenberg M, Chasman DI, Chen YD, Chines PS, Cooper RS, Cucca F, Cusi D, Faire U, Ferrucci L, Franks PW, Froguel P, Gordon-Larsen P, Grabe HJ, Gudnason V, Haiman CA, Hayward C, Hveem K, Johnson AD, Wouter Jukema J, Kardia SLR, Kivimaki M, Kooner JS, Kuh D, Laakso M, Lehtimaki T, Marchand LL, Marz W, McCarthy MI, Metspalu A, Morris AP, Ohlsson C, Palmer LJ, Pasterkamp G, Pedersen O, Peters A, Peters U, Polasek O, Psaty BM, Qi L, Rauramaa R, Smith BH, Sorensen TIA, Strauch K, Tiemeier H, Tremoli E, van der Harst P, Vestergaard H, Vollenweider P, Wareham NJ, Weir DR, Whitfield JB, Wilson JF, Tyrrell J, Frayling TM, Barroso I, Boehnke M, Deloukas P, Fox CS, Hirschhorn JN, Hunter DJ, Spector TD, Strachan DP, van Duijn CM, Heid IM, Mohlke KL, Marchini J, Loos RJF, Kilpelainen TO, Liu CT, Borecki IB, North KE, Cupples LA. Genome-wide meta-analysis of 241,258 adults accounting for smoking behaviour identifies novel loci for obesity traits. Nat Commun. 2017 Apr 26;8:14977. doi: 10.1038/ncomms14977. PMID 28443625
- [Background] 1000 Genomes Project Consortium; Auton A, Brooks LD, Durbin RM, Garrison EP, Kang HM, Korbel JO, Marchini JL, McCarthy S, McVean GA, Abecasis GR. A global reference for human genetic variation. Nature. 2015 Oct 1;526(7571):68-74. doi: 10.1038/nature15393. PMID 26432245
- [Background] McRae AF. Analysis of Genome-Wide Association Data. Methods Mol Biol. 2017;1526:161-173. doi: 10.1007/978-1-4939-6613-4_9. PMID 27896741
- [Background] Purcell S, Neale B, Todd-Brown K, Thomas L, Ferreira MA, Bender D, Maller J, Sklar P, de Bakker PI, Daly MJ, Sham PC. PLINK: a tool set for whole-genome association and population-based linkage analyses. Am J Hum Genet. 2007 Sep;81(3):559-75. doi: 10.1086/519795. Epub 2007 Jul 25. PMID 17701901
- [Background] Team Nutrition. Changing the Scene. Improving the School Nutrition Environment: a Guide to Local Action. Food and Nutrition Service, US Dept of Agriculture; 2000.
- [Background] Gantz W. Food for Thought: Television Food Advertising to Children in the United States. Menlo Park, CA: The Henry J. Kaiser Family Foundation; 2007.
- [Background] Carnell S, Wardle J. Appetitive traits and child obesity: measurement, origins and implications for intervention. Proc Nutr Soc. 2008 Nov;67(4):343-55. doi: 10.1017/S0029665108008641. Epub 2008 Aug 20. PMID 18715519
- [Background] Lohman TG1, Roche AF1, Martorell R1. Anthropometric Standardization Reference Manual. Champaign, IL : Human Kinetics Books; 1988.
- [Background] LeBlanc AG, Katzmarzyk PT, Barreira TV, Broyles ST, Chaput JP, Church TS, Fogelholm M, Harrington DM, Hu G, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tudor-Locke C, Zhao P, Tremblay MS; ISCOLE Research Group. Correlates of Total Sedentary Time and Screen Time in 9-11 Year-Old Children around the World: The International Study of Childhood Obesity, Lifestyle and the Environment. PLoS One. 2015 Jun 11;10(6):e0129622. doi: 10.1371/journal.pone.0129622. eCollection 2015. PMID 26068231
- [Background] Katzmarzyk PT, Barreira TV, Broyles ST, Champagne CM, Chaput JP, Fogelholm M, Hu G, Johnson WD, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Onywera V, Sarmiento OL, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Church TS. The International Study of Childhood Obesity, Lifestyle and the Environment (ISCOLE): design and methods. BMC Public Health. 2013 Sep 30;13:900. doi: 10.1186/1471-2458-13-900. PMID 24079373
- [Background] Mitchell JA, Pate RR, Beets MW, Nader PR. Time spent in sedentary behavior and changes in childhood BMI: a longitudinal study from ages 9 to 15 years. Int J Obes (Lond). 2013 Jan;37(1):54-60. doi: 10.1038/ijo.2012.41. Epub 2012 Mar 20. PMID 22430304
- [Background] Mathie MJ, Coster AC, Lovell NH, Celler BG. Accelerometry: providing an integrated, practical method for long-term, ambulatory monitoring of human movement. Physiol Meas. 2004 Apr;25(2):R1-20. doi: 10.1088/0967-3334/25/2/r01. PMID 15132305
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Petersen AC, Crockett L, Richards M, Boxer A. A self-report measure of pubertal status: Reliability, validity, and initial norms. J Youth Adolesc. 1988 Apr;17(2):117-33. doi: 10.1007/BF01537962. PMID 24277579
- [Background] Carskadon MA, Acebo C. A self-administered rating scale for pubertal development. J Adolesc Health. 1993 May;14(3):190-5. doi: 10.1016/1054-139x(93)90004-9. PMID 8323929
- [Background] Brooks-Gunn J, Warren MP, Rosso J, Gargiulo J. Validity of self-report measures of girls' pubertal status. Child Dev. 1987 Jun;58(3):829-41. PMID 3608653
- [Background] Rideout VJ, Foehr UG, Roberts DF. Generation M2: Media in the Lives of 8- to 18- Year-Olds. Menlo Park, CA; 2010.
- [Background] Marshall TA, Eichenberger Gilmore JM, Broffitt B, Stumbo PJ, Levy SM. Relative validity of the Iowa Fluoride Study targeted nutrient semi-quantitative questionnaire and the block kids' food questionnaire for estimating beverage, calcium, and vitamin D intakes by children. J Am Diet Assoc. 2008 Mar;108(3):465-72. doi: 10.1016/j.jada.2007.12.002. PMID 18313429
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Background] Dixon HG, Scully ML, Wakefield MA, White VM, Crawford DA. The effects of television advertisements for junk food versus nutritious food on children's food attitudes and preferences. Soc Sci Med. 2007 Oct;65(7):1311-23. doi: 10.1016/j.socscimed.2007.05.011. Epub 2007 Jun 22. PMID 17587474
- [Background] Price AL, Patterson NJ, Plenge RM, Weinblatt ME, Shadick NA, Reich D. Principal components analysis corrects for stratification in genome-wide association studies. Nat Genet. 2006 Aug;38(8):904-9. doi: 10.1038/ng1847. Epub 2006 Jul 23. PMID 16862161
- [Background] Wagner DD, Dal Cin S, Sargent JD, Kelley WM, Heatherton TF. Spontaneous action representation in smokers when watching movie characters smoke. J Neurosci. 2011 Jan 19;31(3):894-8. doi: 10.1523/JNEUROSCI.5174-10.2011. PMID 21248113
- [Background] Fischl B, Salat DH, Busa E, Albert M, Dieterich M, Haselgrove C, van der Kouwe A, Killiany R, Kennedy D, Klaveness S, Montillo A, Makris N, Rosen B, Dale AM. Whole brain segmentation: automated labeling of neuroanatomical structures in the human brain. Neuron. 2002 Jan 31;33(3):341-55. doi: 10.1016/s0896-6273(02)00569-x. PMID 11832223
- [Background] Kriegeskorte N, Simmons WK, Bellgowan PS, Baker CI. Circular analysis in systems neuroscience: the dangers of double dipping. Nat Neurosci. 2009 May;12(5):535-40. doi: 10.1038/nn.2303. PMID 19396166
- [Background] Cox RW, Chen G, Glen DR, Reynolds RC, Taylor PA. FMRI Clustering in AFNI: False-Positive Rates Redux. Brain Connect. 2017 Apr;7(3):152-171. doi: 10.1089/brain.2016.0475. PMID 28398812
- [Background] Eklund A, Nichols TE, Knutsson H. Cluster failure: Why fMRI inferences for spatial extent have inflated false-positive rates. Proc Natl Acad Sci U S A. 2016 Jul 12;113(28):7900-5. doi: 10.1073/pnas.1602413113. Epub 2016 Jun 28. PMID 27357684
- [Background] Liang KY, Zeger SL. Longitudinal Data-Analysis Using Generalized Linear-Models. Biometrika. 1986;73(1):13-22. doi:10.1093/biomet/73.1.13.
- [Background] Higgins JP, Whitehead A, Turner RM, Omar RZ, Thompson SG. Meta-analysis of continuous outcome data from individual patients. Stat Med. 2001 Aug 15;20(15):2219-41. doi: 10.1002/sim.918. PMID 11468761
- [Background] Tangney JP, Baumeister RF, Boone AL. High self-control predicts good adjustment, less pathology, better grades, and interpersonal success. J Pers. 2004 Apr;72(2):271-324. doi: 10.1111/j.0022-3506.2004.00263.x. PMID 15016066
- [Background] Kirby KN, Petry NM, Bickel WK. Heroin addicts have higher discount rates for delayed rewards than non-drug-using controls. J Exp Psychol Gen. 1999 Mar;128(1):78-87. doi: 10.1037//0096-3445.128.1.78. PMID 10100392
- [Background] MacKinnon DP. Introduction to Statistical Mediation Analysis. 2008 ed. New York: Lawrene Erlbaum Associates; 2008.
- [Background] MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002 Mar;7(1):83-104. doi: 10.1037/1082-989x.7.1.83. PMID 11928892
- [Background] Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behav Res Methods. 2008 Aug;40(3):879-91. doi: 10.3758/brm.40.3.879. PMID 18697684
- [Background] VanderWeele TJ. Marginal structural models for the estimation of direct and indirect effects. Epidemiology. 2009 Jan;20(1):18-26. doi: 10.1097/EDE.0b013e31818f69ce. PMID 19234398
- [Background] Bollen KA. Structural Equations with Latent Variables. xiv. New York : Wiley; 1989:471-487.
- [Background] Nikolova YS, Ferrell RE, Manuck SB, Hariri AR. Multilocus genetic profile for dopamine signaling predicts ventral striatum reactivity. Neuropsychopharmacology. 2011 Aug;36(9):1940-7. doi: 10.1038/npp.2011.82. Epub 2011 May 18. PMID 21593733
- [Background] Dalley JW, Roiser JP. Dopamine, serotonin and impulsivity. Neuroscience. 2012 Jul 26;215:42-58. doi: 10.1016/j.neuroscience.2012.03.065. Epub 2012 Apr 25. PMID 22542672
- [Background] McClure AC, Tanski SE, Gilbert-Diamond D, Adachi-Mejia AM, Li Z, Li Z, Sargent JD. Receptivity to television fast-food restaurant marketing and obesity among U.S. youth. Am J Prev Med. 2013 Nov;45(5):560-8. doi: 10.1016/j.amepre.2013.06.011. PMID 24139768
- [Background] Fjell AM, Walhovd KB, Brown TT, Kuperman JM, Chung Y, Hagler DJ Jr, Venkatraman V, Roddey JC, Erhart M, McCabe C, Akshoomoff N, Amaral DG, Bloss CS, Libiger O, Darst BF, Schork NJ, Casey BJ, Chang L, Ernst TM, Gruen JR, Kaufmann WE, Kenet T, Frazier J, Murray SS, Sowell ER, van Zijl P, Mostofsky S, Jernigan TL, Dale AM; Pediatric Imaging, Neurocognition, and Genetics Study. Multimodal imaging of the self-regulating developing brain. Proc Natl Acad Sci U S A. 2012 Nov 27;109(48):19620-5. doi: 10.1073/pnas.1208243109. Epub 2012 Nov 12. PMID 23150548
- [Derived] Yeum D, Renier TJ, Carlson DD, Ballarino GA, Lansigan RK, Meyer ML, Loos RJF, Emond JA, Masterson TD, Gilbert-Diamond D. Genetic associations with neural reward responsivity to food cues in children. Front Nutr. 2024 Sep 25;11:1387514. doi: 10.3389/fnut.2024.1387514. eCollection 2024. PMID 39385774